CLINICAL TRIAL: NCT05938881
Title: Long-term Success Rate of Transvaginal Mesh for the Treatment of Pelvic Organ Prolapse: The Extended RCT Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Lan Zhu, Professor, Peking Union Medical College Hospital
Other Study IDs: extended TVM
Record Dates: First submitted 2023-06-28; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; surgery plastic; pelvic floor; polypropylenes
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- self-cut mesh procedure: This procedure is transvaginal mesh implantation surgery for POP patients. Self-cut mesh procedure is an economic pelvic reconstructive surgical operation with use of specially designed puncture needles and self-cut mesh, which mainly provide anterior and apical compartments support, with posterior compartment reinforced by bridge technique repair. The mesh pieces used in this surgery was cut from a single piece of mesh material(TiLOOP 10*15cm) which is much cheaper and readily available. Patients could have transvaginal hysterectomy concomitantly.
  Interventions: Procedure: self-cut mesh procedure
- mesh-kit procedure: This procedure is transvaginal mesh implantation surgery for POP patients.Mesh-kit procedure is refered to pelvic floor reconstructive surgery with titanium-coated meshes kit(TiLOOP TOTAL6).Patients could have transvaginal hysterectomy concomitantly.
  Interventions: Procedure: mesh-kit procedure

INTERVENTIONS:
Procedure: self-cut mesh procedure — transvaginal mesh procedure using self-cut mesh
  Groups: self-cut mesh procedure
Procedure: mesh-kit procedure — transvaginal mesh procedure using mesh-kit
  Groups: mesh-kit procedure

SUMMARY:
The original RCT trial is designed to compare self-tailored titanium-coated polypropylene mesh procedure with mesh-kit in the treatment of POP stage III-IV in terms of efficacy, safety and cost-effective at 1-year follow-up. This study will follow women in the original RCT study for up to 10 years from the time of the surgery to compare success and complication rates in the two groups. Recruitment into this study is open only to women that already participated in previous RCT, no new treatment interventions will be given. Recruitment into the previous RCT is closed. Women will be strongly encouraged to participate in annual examinations and annual telephone surveys but may participate in only one of these study parts if needed.

DETAILED DESCRIPTION:
The previous study is a randomized trial designed to compare the composite success rate between patients with self-cut mesh procedure and those with mesh-kit procedure. The original RCT study includes a 1-year follow up from the time of surgery, which is too short to evaluate the long-term sequelae of the surgical procedures. The goal of this long-term follow-up study is to extend the follow-up of women in the previous RCT study up to 10 years from the time of surgery and to compare the success and complication rates of the two surgical treatment groups over this extended time period.

The primary aim is to determine whether treatment success in women who undergo the above strategies differ at time points through 10 years. A supplemental study investigates the long-term success rate and complications of transvaginal mesh procedure in women in both of the study arms.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in previous RCT study

Exclusion Criteria:

* Inability to provide informed consent. Informed consent will be obtained prior to each telephone interview and each in-person visit.
* Subjects who appear to have cognitive deficits during the in-person visit or site telephone interview will be withdrawn from the study by the study coordinator.

Ages: 53 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All women enrolled in previous RCT study are invited to this extended study.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2033-01-12 (Estimated); Study Completion 2033-03-12 (Estimated)

PRIMARY OUTCOMES:
Composite success | up to 10 years after procedure
  To determine the long-term (up to 10 years) composite success rate of both procedure (defined as leading edge above the hymen (i.e Ba, C, Bp<0 cm) AND deny vaginal bulging symptoms indicated by a negative response question 3 of the pelvic floor distress inventory- 20 (PFDI-20): "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area? AND no re-operation or pessary treatment for POP), and whether composite success rate differs between women who had self-cut mesh procedure vs. those who had mesh-kit procedure; This outcome measure is cumulative across the original RCT trial and continued through the extended trial follow-up with non-failures tracked either until failure or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)

SECONDARY OUTCOMES:
anatomic outcomes | up to 10 years after operation
  Anatomic failure was defined as POPQ system leading edge at or beyond the hymen (i.e Ba, C, Bp≥0 cm). This outcome measure is cumulative across the original RCT trial and continued through the extended follow-up study with non-failures tracked either until failure or until study completion/dropping out of the study (lost to follow-up, withdrawal, etc.)
Change From Baseline PFIQ-7 Score | up to 10 years after operation
  The Pelvic Floor Impact Questionnaire measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of 3 scales: the Urinary Impact Questionnaire (UIQ; 4 subscales, range 0-400), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; 4 subscales, range 0-400), and the Colorectal-Anal Impact Questionnaire (CRAIQ; 4 subscales, range 0-400). Scores are calculated by multiplying the mean value of all answered questions for a subscale by 100 divided by 3. The subscales are then added together. The range of responses is: 0-400 with 0 (least negative impact) to 400 (most negative impact). Change = (Year [up to 10 years] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Change From Baseline PFDI-20 Score | up to 10 years after operation
  The Pelvic Floor Distress Inventory is a validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of 3 scales: 1. Pelvic Organ Prolapse Distress Inventory (with 3 subscales), 2. Colorectal Anal Distress Inventory (with 4 subscales), and 3. Urinary Distress Inventory (with 3 subscales). Scores are calculated by multiplying the mean value of all questions answered by 25 for the subscales and then adding the subscales. The range of responses for the CRADI is: 0-400 with 0 (least distress) to 400 (most distress). Change = (Year [up to 10 years] Score - Baseline Score). Lower scores indicate better function / fewer symptoms.
Change From Baseline PISQ-12 Score | up to 10 years after operation
  The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, (PISQ-12) is a questionnaire measuring the impact of POP symptoms on sexual function and satisfaction. The PISQ-12 Score ranges from 0 to 48 with higher scores indicating better function/satisfaction. Change = (Year [up to 10 years] Score - Baseline Score). Higher scores indicate better function / fewer symptoms.
Symptomatic improvement using patient global impression of change (PGI-C) | up to 10 years after operation
  The Patient Global Impression of Change (PGI-C) is a patient-reported measure of perceived change with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better).
Complications | up to 10 years after operation
  Using IUGA/ICS Joint Terminology CTS coding system and Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Foshan Maternal and Child Health Care Hospital, Foshan, Guangdong
  - The First Affiliated Hospital of Guangdong Medical College, Guangzhou, Guangdong
  - Changsha Maternal and Child Health Care Hospital, Changsha, Hunan
  - The Secong Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Maternal and Child Health Care Hospital, Wuxi, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanxi Provincial People's Hosptial, Xi’an, Shanxi
  - Sichuan University West China Second University Hospital, Chengdu, Sichuan
  - the First Affiliated Hosptial of Xinjiang Medical University, Ürümqi, Xiangjiang
  - The People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Peking Union Medical College Hospital, Beijing